CLINICAL TRIAL: NCT06187168
Title: Intra-operative Hypotension and Sepsis After Endoscopic Retrograde Cholangiopancreatography: A Prospective Cohort Study
Brief Title: Risk Factors of Post-ERCP Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: R.23.11.2387
Record Dates: First submitted 2023-12-17; First posted 2024-01-02 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Sepsis; Intraoperative Hypotension; Bacteremia Sepsis
MeSH Terms: conditions — Sepsis | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- intraoperative hypotension: The exposure is intra-operative hypotension during the ERCP procedure (hypotension is defined as a 20% reduction in the mean arterial blood pressure (MAP) or systolic arterial blood pressure (SAP) < 90 mmHg during CBD manipulation or after obstruction relief). The basal blood pressure (BP) will be the immediate reading before the endoscope insertion while the patient is in his left lateral position.
  Interventions: Procedure: exposure to hypotension during the Endoscopic Retrograde Cholangiopancreatography (ERCP) for obstructive jundice.
- No intraoperative hypotension: Not meeting the above definition of hypotension per our protocol (by timing, threshold, and method).

INTERVENTIONS:
Procedure: exposure to hypotension during the Endoscopic Retrograde Cholangiopancreatography (ERCP) for obstructive jundice. — This is not an intended intervention in the study. This cohort study will study the exposure to intraoperative hypotension and the occurrence of sepsis after the ERCP procedures.
  Groups: intraoperative hypotension

SUMMARY:
For the treatment of numerous biliary and pancreatic problems, the procedure known as endoscopic retrograde cholangiopancreatography (ERCP) is regarded as a crucial therapeutic intervention. However, ERCP is known to be connected to a variety of issues, including post-ERCP sepsis. This study's goal is to investigate the relationship between unexplained hypotension during or just after surgery and the emergence of sepsis after ERCP.

DETAILED DESCRIPTION:
At the Gastrointestinal Surgery Centre, Mansura University, Egypt, a cohort study will be conducted on a sample of 50 adult (18+) patients who undergoing ERCP. Hypotension that occurred during surgery or shortly after will be classified as exposure when it cannot be linked to a particular cause. In this study, post-ERCP sepsis will be the major outcome measure, while other ERCP-related sequelae will be the supplementary outcome measures.

Discussion:

The findings of this study will significantly advance our understanding of the potential link between intraoperative hypotension and the development of post-ERCP sepsis. This study's goal is to increase knowledge of the challenges presented by ERCP, which will aid in the creation of patient treatment methods that are more effective.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing ERCP for obstructive jaundice
* Adult (Older than 18 years old)
* Written Informed Consent

Exclusion Criteria:

* Already on sepsis before the ERCP
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will include 100 adult patients (≥ 18years) undergoing ERCP for obstructive jaundice at the GISC during the study period for obstructive jaundice.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-23 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Post-ERCP Sepsis | 24 hours after ERCP
  Definition: SOFA score ≥ 2 or increase in the SOFA score by ≥ 2 from the baseline SOFA score ≥ 2 or increase in the SOFA score by ≥ 2 from the baseline (dicotomus outcome: yes or no)

SECONDARY OUTCOMES:
Hospital readmission | 30 days after ERCP
  Hospital readmission (dicotomus outcome: yes or no)
Post-ERCP ICU admission | 7 days after ERCP
  post-ERCP admission to the ICU for any cause (dicotomus outcome: yes or no)
Length of hospital stay | 30 days after ERCP
  in days (continuous outcome)
Postoperative bacteremia | 24 hours after surgery
  Bactermia on blood culture (post-ERCP in comparison to the pre-ERCP blood culture): (dicotomus outcome: yes or no)
Post-ERCP pancreatitis | 24 hours after ERCP
  Raised lipases and amylase (dicotomus outcome: yes or no)
Post-ERCP RBCs transfusion | 24 hours after ERCP
  any amount of red blood tranfusion after the ERCP (dicotomus outcome: yes or no)
30-day all-cause mortality | 30 days after ERCP
  Death of any cause (dicotomus outcome: yes or no)
Delayed post-ERCP Sepsis | 7 days after ERCP procedure
  SOFA score ≥ 2 or increase in the SOFA score by ≥ 2 from the baseline (dicotomus outcome: yes or no)

CONTACTS AND LOCATIONS:
Overall Officials: Moataz M Emara, MD, EDAIC, Study Chair — Mansoura University Hospital
Locations (1):
- Mansoura Univesity Faculty of Medicine, Al Mansurah, Aldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The anonymized patient data will be available with the principal investigator and can be shared on reasonable request after approval of the IRB.
Time Frame: within 2 years after publication
Access Criteria: with contact with the principal investigator with reasonable request and approval of the local IRB.